CLINICAL TRIAL: NCT06299449
Title: Clinical and Radiographic Outcomes of Computer Guided Immediate Implant Placement Utilizing Artificial Intelligence Assisted Socket Shield Approach: Randomized Clinical Trial
Brief Title: Artificial Intelligence Assisted Socket Shield With Computer Guided Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, Assistant Professor of periodontology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-174
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Implant Complication; Dental Implant Failed

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): conventional socket shield with conventional simultaneous implant placement
  Interventions: Procedure: free-hand socket shield
- study group (Experimental): computer guided implant placement combined with artificial intelligence-assisted socket shield.
  Interventions: Procedure: AI/guided socket shield

INTERVENTIONS:
Procedure: free-hand socket shield — Immediate Implant Placement Using Socket Shield Technique with autogenous whole tooth graft after immediate implantation using Socket Shield Technique, the palatal root portion and the decoronated crown will be converted to autogenous whole tooth graft and used for grafting the defect between the socket shield and the implant fixture
  Other Names: Elamrousy Novel Approach of Socket Shield Technique
  Arms: control group
Procedure: AI/guided socket shield — The patient specific guides will be placed at the pre-planned positions at the labial buccal mucosa.
  using artificial intelligence the socket shield approach will be planned to keep the buccal shield and using surgical guide the shield will be preciesly prepared followed by guided implant placement and whole tooth grafting of the jumping gap
  Other Names: AI/guided Elamrousy Novel Approach of Socket Shield Technique
  Arms: study group

SUMMARY:
Aim of the current randomized clinical trial is to evaluate and compare the effectiveness of computer-guided immediate implant placement performed simultaneously with artificial intelligence assisted socket shield technique versus conventional approach.

DETAILED DESCRIPTION:
Guided implant surgery was used in dental implant surgery to achieve accuracy and an overall predictability. Successful guided implant workflow depends on 3-dimensional image acquisition and precise model fabrication.

Artificial intelligence application in implant dentistry has ushered in a new era of precision and efficiency demonstrating improved implant survival rates and patient satisfaction and enhance the integration of technologies with digital workflows.

ELIGIBILITY:
Inclusion Criteria:

* above the age of 18years
* presence of non-restorable maxillary anterior tooth
* had intact socket walls following tooth extraction
* the gingival biotype was thick.

Exclusion Criteria:

* history of systemic condition
* history of using bisphosphonates or other drugs that might impact bone turnover
* a history of smoking during the previous five years,
* a history of any acute infections at the surgical site,
* teeth having root resorptions

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-10-26 (Actual)

PRIMARY OUTCOMES:
Stability Quotient of dental implant | 9-month.
  Osstell TM was used to record the primary stability.ISQ, or Implant Stability Quotient, is a scale from 1 to 100 and is a measure of the stability of an implant. The ISQ scale has a non-linear correlation to micro mobility. With more than 1400 scientific references, investigators now know that high stability means >70 ISQ, between 60-69 is medium stability and < 60 ISQ is considered as low stability
pink esthetic score | 9-month.
  The pink esthetic score (PES) evaluates the esthetic outcome of soft tissue around implant-supported single crowns in the anterior zone by awarding seven points for the mesial and distal papilla, soft-tissue level, soft-tissue contour, soft-tissue color, soft-tissue texture, and alveolar process deficiency.Using a 0-1-2 scoring system, 0 being the lowest, 2 being the highest value, the maximum achievable PES was 14
Midfacial Mucosal Alterations | 9-month.
  digital intraoral scans were recorded. To quantify the vertical changes in the soft tissues around implants buccally, the collected scans were digitally superimposed via matching Gom inspect software
facial marginal bone level | 9-month
  Utilizing CBCT sagittal sections, the BMBL was evaluated by computerized analysis. Navigation was done on the multiplanar display until the implant's precise same-view location was established on the reformatted cross-sectional section and panoramic view.

CONTACTS AND LOCATIONS:
Overall Officials: Walid AH Elamrousy, PhD, Study Director — Faculty of Oral and Dental Medicine, Kafrelsheikh University
Locations (1):
- faculty of dentistry, kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No
the new approach of using artificial intelligence to assist in the planning of socket shield technique will not be shared